CLINICAL TRIAL: NCT06767345
Title: Comparing the Moderate Intensity STatin With Ezetimibe COmbination TheraPy With High Intensity Statin Monotherapy on Coronary PLAQUE Stabilization
Brief Title: Comparison of Moderate-Intensity Statin Plus Ezetimibe vs. High-Intensity Statin for Coronary Plaque Stabilization
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Korea University Anam Hospital (Other)
Collaborators: Yuhan Corporation (Industry); Hanmi Pharmaceutical co., ltd. (Other)
Responsible Party: Principal Investigator, Soon Jun Hong, Professor, Korea University Anam Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STOP-PLAQUE
Record Dates: First submitted 2025-01-03; First posted 2025-01-09 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Coronary Artery Disease; Atherosclerosis of Coronary Artery; Plaque, Atherosclerotic
MeSH Terms: conditions — Coronary Artery Disease; Plaque, Atherosclerotic | interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors; Ezetimibe; Combined Modality Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High Intensity Statin monotherapy (Active Comparator): Rosuvastatin 20mg once a daily
  Interventions: Drug: statins, ezetimibe
- Combination therapy (Experimental): Rosuvastatin 10mg plus Ezetimibe 10mg fixed dose single-pill combination
  Interventions: Drug: Combination therapy

INTERVENTIONS:
Drug: statins, ezetimibe — Rosuvastatin 20mg once daily
  Arms: High Intensity Statin monotherapy
Drug: Combination therapy — Rosuvastatin 10mg + Ezetimibe 10mg
  Arms: Combination therapy

SUMMARY:
This study is a prospective, multicenter, randomized clinical trial aimed at comparing the effects of moderate-intensity statin plus ezetimibe combination therapy versus high-intensity statin monotherapy on coronary plaque stabilization. Using advanced imaging techniques such as near-infrared spectroscopy-intravascular ultrasound (NIRS-IVUS), the trial evaluates whether the combination therapy is non-inferior to monotherapy in stabilizing coronary plaques over 52 weeks. The primary endpoint is the percentage change in coronary atheroma volume (PAV) assessed by grayscale IVUS, with secondary outcomes including changes in lipid core burden, inflammatory markers, and clinical events like myocardial infarction and ischemic stroke. The study plans to enroll 408 patients undergoing coronary intervention across 7 domestic institutions, with rigorous follow-up protocols and adherence to international research guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women over the age of 18 years.
* Patients with coronary artery disease undergoing a coronary intervention procedure using intravascular imaging.
* At least one major native coronary artery ("target vessel") meeting all the following criteria for intracoronary imaging immediately following a qualifying PCI procedure:

  * Angiographic evidence of coronary artery stenosis ≥30% by angiographic visual estimation.
  * Target vessel is accessible to the imaging catheter and suitable for intracoronary imaging in the proximal 50 mm segment.
  * Target vessel is not a bypass graft (aortic or arterial) or a bypassed graft vessel.
  * Target vessel has not undergone PCI within the target segment.
  * Target vessel is not a candidate for PCI at the time of the procedure or for 6 months thereafter (per investigator's judgment).
* Patients who have provided written informed consent to participate in the study.

Exclusion Criteria:

* Left main stem lesion: Left main coronary artery stenosis ≥50% by coronary angiographic visual estimation.
* History of coronary artery bypass graft surgery (CABG).
* Unstable clinical condition (hemodynamic or electrical instability).
* Severe coronary artery calcification or tortuosity interfering with IVUS, NIRS, or evaluation.
* Uncontrolled cardiac arrhythmia (recurrent and symptomatic ventricular tachycardia or atrial fibrillation with rapid ventricular response) not controlled by medication within 3 months prior to screening.
* Active liver disease or liver dysfunction.
* Severe renal dysfunction (eGFR <30 mL/min/1.73m²)
* Known allergy to contrast media, heparin, aspirin, ticagrelor, or prasugrel.
* Active infection or major hematologic, metabolic, or endocrine dysfunction as determined by the investigator.
* Planned surgery within 12 months.
* Currently enrolled in another investigational device or drug study.
* Estimated life expectancy of less than 2 years.
* Women of childbearing potential (under 50 years of age) who:

  * Had their last menstrual period within the last 12 months.
  * Have not had tubal ligation, oophorectomy, or hysterectomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 408 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2028-01-25 (Estimated); Study Completion 2028-06-25 (Estimated)

PRIMARY OUTCOMES:
percentage change in coronary atheroma volume (PAV) by gray-scale IVUS from baseline to week 52. | 52 weeks

SECONDARY OUTCOMES:
Change from baseline to week 52 in total lipid core BMI measured by NIRS (LCBItotal) | 52 weeks
Change in maximum LCBI within a 4-mm bin measured by NIRS from baseline to week 52 (maxLCBI4mm) | 52 weeks
Change in corrected total atherosclerotic plaque volume (NTAV) measured by IVUS from baseline to week 52 | 52 weeks

OTHER OUTCOMES:
Changes in LDL-cholesterol from baseline to 52 weeks and associations with plaque progression/regression indices | 52 weeks
  LDL-cholesterol levels measured in mg/dL using [specific lab assay name]. Blood samples will be collected at baseline and after 52 weeks.
All deaths from baseline to week 52 | 52 weeks
Cardiac-related deaths from baseline to week 52 | 52 weeks
Nonfatal myocardial infarction from baseline to week 52 | 52 weeks
Ischemic Coronary Revascularization From Baseline to Week 52 | 52 weeks
Ischemic Stroke/TIA from Baseline to Week 52 | 52 weeks
Incidence of new diabetes from baseline to week 52 | 52 weeks
Incidence of statin-associated muscle syndrome (SAMS) from baseline to week 52 | 52 weeks
Adherence from baseline to week 52 (80% or greater) | 52 weeks
  Proportion of patients achieving ≥80% adherence to prescribed medication from baseline to week 52
Cataract incidence from baseline to 52 weeks | 52 weeks
Changes in hsCRP from baseline to 52 weeks and associations with plaque progression/regression indices | 52 weeks
Changes in hsTnT from baseline to 52 weeks and associations with plaque progression/regression indices | 52 weeks
Changes in NT-pro-BNP from baseline to 52 weeks and associations with plaque progression/regression indices | 52 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Anam Hospital, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Preiss D, Seshasai SR, Welsh P, Murphy SA, Ho JE, Waters DD, DeMicco DA, Barter P, Cannon CP, Sabatine MS, Braunwald E, Kastelein JJ, de Lemos JA, Blazing MA, Pedersen TR, Tikkanen MJ, Sattar N, Ray KK. Risk of incident diabetes with intensive-dose compared with moderate-dose statin therapy: a meta-analysis. JAMA. 2011 Jun 22;305(24):2556-64. doi: 10.1001/jama.2011.860. PMID 21693744
- [Background] Sattar N, Preiss D, Murray HM, Welsh P, Buckley BM, de Craen AJ, Seshasai SR, McMurray JJ, Freeman DJ, Jukema JW, Macfarlane PW, Packard CJ, Stott DJ, Westendorp RG, Shepherd J, Davis BR, Pressel SL, Marchioli R, Marfisi RM, Maggioni AP, Tavazzi L, Tognoni G, Kjekshus J, Pedersen TR, Cook TJ, Gotto AM, Clearfield MB, Downs JR, Nakamura H, Ohashi Y, Mizuno K, Ray KK, Ford I. Statins and risk of incident diabetes: a collaborative meta-analysis of randomised statin trials. Lancet. 2010 Feb 27;375(9716):735-42. doi: 10.1016/S0140-6736(09)61965-6. Epub 2010 Feb 16. PMID 20167359
- [Background] Davis JW, Weller SC. Intensity of statin therapy and muscle symptoms: a network meta-analysis of 153 000 patients. BMJ Open. 2021 Jun 15;11(6):e043714. doi: 10.1136/bmjopen-2020-043714. PMID 34130955
- [Background] Maron DJ, Hochman JS, Reynolds HR, Bangalore S, O'Brien SM, Boden WE, Chaitman BR, Senior R, Lopez-Sendon J, Alexander KP, Lopes RD, Shaw LJ, Berger JS, Newman JD, Sidhu MS, Goodman SG, Ruzyllo W, Gosselin G, Maggioni AP, White HD, Bhargava B, Min JK, Mancini GBJ, Berman DS, Picard MH, Kwong RY, Ali ZA, Mark DB, Spertus JA, Krishnan MN, Elghamaz A, Moorthy N, Hueb WA, Demkow M, Mavromatis K, Bockeria O, Peteiro J, Miller TD, Szwed H, Doerr R, Keltai M, Selvanayagam JB, Steg PG, Held C, Kohsaka S, Mavromichalis S, Kirby R, Jeffries NO, Harrell FE Jr, Rockhold FW, Broderick S, Ferguson TB Jr, Williams DO, Harrington RA, Stone GW, Rosenberg Y; ISCHEMIA Research Group. Initial Invasive or Conservative Strategy for Stable Coronary Disease. N Engl J Med. 2020 Apr 9;382(15):1395-1407. doi: 10.1056/NEJMoa1915922. Epub 2020 Mar 30. PMID 32227755
- [Background] Park SJ, Ahn JM, Kang DY, Yun SC, Ahn YK, Kim WJ, Nam CW, Jeong JO, Chae IH, Shiomi H, Kao HL, Hahn JY, Her SH, Lee BK, Ahn TH, Chang KY, Chae JK, Smyth D, Mintz GS, Stone GW, Park DW; PREVENT Investigators. Preventive percutaneous coronary intervention versus optimal medical therapy alone for the treatment of vulnerable atherosclerotic coronary plaques (PREVENT): a multicentre, open-label, randomised controlled trial. Lancet. 2024 May 4;403(10438):1753-1765. doi: 10.1016/S0140-6736(24)00413-6. Epub 2024 Apr 8. PMID 38604213
- [Background] Kim BK, Hong SJ, Lee YJ, Hong SJ, Yun KH, Hong BK, Heo JH, Rha SW, Cho YH, Lee SJ, Ahn CM, Kim JS, Ko YG, Choi D, Jang Y, Hong MK; RACING investigators. Long-term efficacy and safety of moderate-intensity statin with ezetimibe combination therapy versus high-intensity statin monotherapy in patients with atherosclerotic cardiovascular disease (RACING): a randomised, open-label, non-inferiority trial. Lancet. 2022 Jul 30;400(10349):380-390. doi: 10.1016/S0140-6736(22)00916-3. Epub 2022 Jul 18. PMID 35863366
- [Background] Raber L, Ueki Y, Otsuka T, Losdat S, Haner JD, Lonborg J, Fahrni G, Iglesias JF, van Geuns RJ, Ondracek AS, Radu Juul Jensen MD, Zanchin C, Stortecky S, Spirk D, Siontis GCM, Saleh L, Matter CM, Daemen J, Mach F, Heg D, Windecker S, Engstrom T, Lang IM, Koskinas KC; PACMAN-AMI collaborators. Effect of Alirocumab Added to High-Intensity Statin Therapy on Coronary Atherosclerosis in Patients With Acute Myocardial Infarction: The PACMAN-AMI Randomized Clinical Trial. JAMA. 2022 May 10;327(18):1771-1781. doi: 10.1001/jama.2022.5218. PMID 35368058